CLINICAL TRIAL: NCT07063368
Title: Combined Effects of Otago Exercises and Systematic Desensitization on Balance,Fall Risk and Basophobia Among Post Stroke Older Adults
Brief Title: Effects of Otago Exercises and Systematic Desensitization on Balance,Fall Risk and Basophobia Among Post Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0254
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Fall Risk; Otago exercises; Balance; Systematic desensitization; Basophobia
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Otago Exercises and systematic desensitization with routine physical therapy (Experimental): Group A emphasizes a combination of Otago exercises and systematic desensitization alongside routine physical therapy. The session begins with a 5-minute warm-up, followed by 7 minutes of Otago balance exercises and 8 minutes of Otago strength exercises. This is complemented by 15 minutes of routine physical therapy focusing on strength and mobility, 5 minutes of flexibility and stretching, and 7 minutes dedicated to relaxation training. The session concludes with 10 minutes of gradual exposure and visualization exercises, allowing participants to mentally navigate safe environments and mildly fear-inducing situations, followed by a 3-minute discussion and feedback segment.
  Interventions: Other: Otago exercises and systematic desensitization with routine physical therapy
- Otago Exercises and Routine Physical Therapy (Experimental): Group B, centers solely on Otago exercises integrated with routine physical therapy. This group starts with a 10-minute warm-up, followed by 10 minutes of Otago balance exercises and another 10 minutes for Otago strength exercises. The session continues with 20 minutes of routine physical therapy focused on strength and mobility, concluding with 10 minutes dedicated to flexibility and stretching exercises.
  Interventions: Other: Otago Exercises and Routine physical Therapy
- Systematic desensitization and Routine physical therapy (Experimental): Group C combines systematic desensitization with routine physical therapy. The session begins with a 5-minute warm-up, followed by 20 minutes of strength and mobility exercises, and 5 minutes of flexibility and stretching. Participants then engage in 10 minutes of relaxation training, which includes reviewing goals and practicing deep breathing exercises. The session further incorporates 15 minutes of gradual exposure and visualization, allowing participants to confront their fears in a controlled manner, and wraps up with a 5-minute discussion and feedback period.
  Interventions: Other: Systematic desensitization and routine physical therapy

INTERVENTIONS:
Other: Otago exercises and systematic desensitization with routine physical therapy — Warm-up (5 minutes) Marching in place (assisted), arm swings, side steps Otago Balance Exercises (7 minutes) Knee bends (with support), heel-to-toe stand (with support), side hip abduction (with support) Otago Strength Exercises (8 minutes) Ankle dorsiflexion, seated knee extensions, seated marching Routine Physical Therapy - Strength and Mobility Exercises (15 minutes) Assisted squats or sit-to-stand exercises, standing calf raises (with support), seated bicep curls, seated shoulder press Routine Physical Therapy - Flexibility and Stretching (5 minutes) Hamstring, quadriceps, shoulder, and neck stretches Relaxation Training (7 minutes) Review goals, PMR, deep breathing exercises Gradual Exposure and Visualization (10 minutes) Visualization of safe environments, standing up, walking on flat surfaces, and mildly fear-inducing situations (with assistance) Discussion and Feedback (3 minutes) Share experiences, provide feedback, assign homework
  Arms: Otago Exercises and systematic desensitization with routine physical therapy
Other: Otago Exercises and Routine physical Therapy — Warm-up (10 minutes) Marching in place, arm swings, and side steps. Otago Balance Exercises (10 minutes) Knee bends, heel-to-toe stand, side hip abduction. Otago Strength Exercises (10 minutes) Ankle dorsiflexion, seated knee extensions, seated marching. Routine Physical Therapy - Strength and Mobility Exercises (20 minutes) Assisted squats or sit-to-stand exercises, standing calf raises with support, seated bicep curls, seated shoulder press.
  Routine Physical Therapy - Flexibility and Stretching (10 minutes) Hamstring stretch, quadriceps stretch, shoulder and neck stretches, seated torso twist.
  Arms: Otago Exercises and Routine Physical Therapy
Other: Systematic desensitization and routine physical therapy — Warm-up (5 minutes) Marching in place, arm swings, and side steps. Routine Physical Therapy - Strength and Mobility Exercises (20 minutes) Assisted squats or sit-to-stand exercises, standing calf raises with support, seated bicep curls, seated shoulder press.
  Routine Physical Therapy - Flexibility and Stretching (5 minutes) Hamstring stretch, quadriceps stretch, shoulder and neck stretches. Relaxation Training (10 minutes) Review goals and expectations, PMR, deep breathing exercises. Gradual Exposure and Visualization (15 minutes) Visualization of safe environments, standing up, walking on flat surfaces, and mildly fear-inducing situations (with assistance).
  Discussion and Feedback (5 minutes) Share experiences, provide feedback, and assign homework.
  Arms: Systematic desensitization and Routine physical therapy

SUMMARY:
The aim of the study is to determine the combined effects of Otago exercises and systematic desensitization on balance, fall risk, and basophobia among post-stroke older adults.

DETAILED DESCRIPTION:
Stroke survivors often face challenges such as impaired balance, heightened fall risk, and basophobia (fear of falling), which significantly impact their daily lives and rehabilitation outcomes. Stroke patients have a two-fold higher risk of falling than other patients of the same age or gender.In particular, 30% to 50% of the elderly those over 65 years old, experience falls every year. The Otago Exercise Program, recognized for its efficacy in improving balance and reducing falls among older adults, and systematic desensitization, a psychological intervention aimed at reducing fear and anxiety related to falling, offer complementary approaches to address these challenges. This study aims to investigate the combined effects of Otago exercises and systematic desensitization on balance, fall risk, and basophobia among post-stroke older adults.

This randomized controlled trial will be conducted at Allama Iqbal Memorial Teaching Hospital Sialkot over six months. The sample size will consist of 51 participants. Participants who meet the inclusion criteria will be taken through a non-probability convenience sampling technique, which will further be randomized through flip coin method. 17 Participants will be assigned to group A (otago exercise, systematic desensitization and routine physical therapy, 17 participants to group B( Otago Exercises and Routine Physical therapy ) and 17 participants were included in group C ( Systematic desensitization and Routine physical therapy only ).

Data will be collected using various assessment tools, including the Berg Balance Scale to assess balance , Timed up and go test for dynamic balance, Functional Reach Test for static balance, Fall Risk assessment scale to assess risk of fall, Fall Efficacy Scale International for risk of fall, and Fear of fall avoidance behavior questionnaire for basophobia. Pre-intervention assessments will be conducted for all three groups. The effects of the interventions will be measured at pre-treatment, 4th week, and post-intervention. Data analysis will be performed by using SPSS 26 software.

ELIGIBILITY:
Inclusion Criteria :

* Both male and female patients
* 40 to 70 Years of age
* sub-acute ischemic stroke
* Ability to walk with or without a caregiver
* No cognitive dysfunction that would hinder understanding of the instructions
* MoCA score between 18-24

Exclusion Criteria :

* Patients previous participation in studies similar to the present study.
* Participants who have other medical conditions such as severe arthritis or joint injuries.
* Participants who have a history of significant neurological or psychiatric disorders
* Participants who have severe visual or hearing impairments
* Participants who are currently participating in another clinical trial or research study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Fall Risk Assessment Scale | 8 weeks
  It is a 4-item falls-risk screening tool for sub-acute and residential care. The FRAT has three sections: Part 1 - Fall Risks, Part 2 -Risk factor checklist, Part 3 :Action Plan. A score of 0 to 5 indicates a low risk of falling, a score of 6 to 20 a medium risk, and a score 21 to 45 a high risk.
Fall Efficacy Scale International | 8 weeks
  The Falls Efficacy Scale International (FES-I) is a measure of fear of falling. It is a 16 item questionnaire, useful to the researchers and clinicians interested in fear of falling, with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).
Berg Balance Scale | 8 weeks
  The Berg Balance Scale (BBS) is a clinical tool used to assess balance and risk of falling. It consists of 14 simple tasks, such as standing, sitting, and reaching, each scored on a scale of 0 to 4. The total score helps determine the level of balance impairment.

SECONDARY OUTCOMES:
Timed Up and Go test | 8 weeks
  The Timed Up and Go (TUG) test is a simple and quick assessment used to evaluate a person's mobility, balance, walking ability, and fall risk. It involves timing an individual as they stand up from a chair, walk three meters, turn around, walk back, and sit down. A time of 12 seconds or more typically indicates a higher risk of falling
Functional Reach Test | 8 weeks
  It is a quick, single-task, dynamic test that is used to predicting falls in older adults. This test measures the margin of stability along with the ability to measure balance during a functional task.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Jabeen, PhD, Principal Investigator — Riphah International University
Locations (1):
- Allama Iqbal Memorial Teaching Hospiatl, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peng Y, Wang Y, Zhang L, Zhang Y, Sha L, Dong J, He Y. Virtual reality exergames for improving physical function, cognition and depression among older nursing home residents: A systematic review and meta-analysis. Geriatr Nurs. 2024 May-Jun;57:31-44. doi: 10.1016/j.gerinurse.2024.02.032. Epub 2024 Mar 18. PMID 38503146
- [Background] Wang J, Li Y, Yang GY, Jin K. Age-Related Dysfunction in Balance: A Comprehensive Review of Causes, Consequences, and Interventions. Aging Dis. 2024 Jan 24;16(2):714-737. doi: 10.14336/AD.2024.0124-1. PMID 38607735
- [Background] Zhong YJ, Meng Q, Su CH. Mechanism-Driven Strategies for Reducing Fall Risk in the Elderly: A Multidisciplinary Review of Exercise Interventions. Healthcare (Basel). 2024 Nov 29;12(23):2394. doi: 10.3390/healthcare12232394. PMID 39685016
- [Background] Yi M, Zhang W, Zhang X, Zhou J, Wang Z. The effectiveness of Otago exercise program in older adults with frailty or pre-frailty: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2023 Nov;114:105083. doi: 10.1016/j.archger.2023.105083. Epub 2023 Jun 22. PMID 37390692
- [Background] Chiu HL, Yeh TT, Lo YT, Liang PJ, Lee SC. The effects of the Otago Exercise Programme on actual and perceived balance in older adults: A meta-analysis. PLoS One. 2021 Aug 6;16(8):e0255780. doi: 10.1371/journal.pone.0255780. eCollection 2021. PMID 34358276
- [Background] Yang Y, Wang K, Liu H, Qu J, Wang Y, Chen P, Zhang T, Luo J. The impact of Otago exercise programme on the prevention of falls in older adult: A systematic review. Front Public Health. 2022 Oct 20;10:953593. doi: 10.3389/fpubh.2022.953593. eCollection 2022. PMID 36339194